CLINICAL TRIAL: NCT01325090
Title: Early Administration of Botulinum Toxin Type A (Botox®) in Neuropathic Pain Due to Thoracoscopy or Thoracotomy: a Randomized, Double Blind, Placebo Controlled Study
Brief Title: Early Administration of Botox® in Neuropathic Pain Due to Thoracoscopy or Thoracotomy
Acronym: APTODON
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: I09006 / APTODON; 2010-021506-38 (EudraCT Number)
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2011-03

CONDITIONS: Pain Due to Certain Specified Procedures; Neuropathic Pain
Keywords: neuropathic pain due to thoracotomy; Neuropathic Pain Due to Thoracoscopy
MeSH Terms: conditions — Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOTOX (Experimental): Patients will receive in one session multiple intradermal injections of Botox, in order to cover the whole painful area
  Interventions: Drug: BOTOX
- PLACEBO (Placebo Comparator): Patients will receive in one session multiple intradermal injections of placebo , in order to cover the whole painful area
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: BOTOX — A syringe of 1 ml contain 25 Allergan units.
  Arms: BOTOX
Other: PLACEBO — The pharmacist will fill syringes in tuberculins of 1 ml with injectable solution of sodium chloride of 0,9 %.
  Arms: PLACEBO

SUMMARY:
Botulinum toxin type A has been reported to inhibit the release of various pain neurotransmitters (SP, CGRP, glutamate) responsible for neurogenic inflammation, a process that results from the sensitization of C-fiber nociceptors (peripheral sensitization). This action is probably responsible for the analgesic effect of botulinum toxin type A recently demonstrated in patients with neuropathic pain of peripheral origin.In those studies, patients had been suffering for years. The investigators can hypothesizes that earlier administration of Botox in the course of neuropathic pain might prevent central sensitization, that is secondary to peripheral sensitization. The investigators can hope to increase efficacy of Botulinum toxin type A injections and to prevent chronification of pain.

ELIGIBILITY:
Inclusion Criteria:

* daily pain, for 3 months, secondary to thoracoscopy or thoracotomy, of neuropathic origin (DN4 questionary)

Exclusion Criteria:

* contraindications for botulinum toxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
decrease in average pain intensity as measured by the Brief Pain Inventory (BPI) | one month

SECONDARY OUTCOMES:
VAS in the last 24 hours | 24 hours
Neuropathic Pain Inventory | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Danièle RANOUX, MD, Principal Investigator — University Hospital, Limoges